CLINICAL TRIAL: NCT04297501
Title: Effect of 1-year Antiretroviral Treatment on Gut Microbiota Diversity and Composition in Treatment-naïve HIV-infected Chinese Individuals
Brief Title: Gut Microbiota Changes of HIV Patients Before and After One Year of ART
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CACTGUT18A
Record Dates: First submitted 2018-06-08; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2018-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Facal samples were collected and then DNA was retracted, all samples were stored in -80oC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All enrolled participants in this study
  Interventions: Drug: Antiretroviral Therapy

INTERVENTIONS:
Drug: Antiretroviral Therapy — All participants receive antiretroviral therapy to control virus replication and restore CD4+ T-cell count.

SUMMARY:
HIV infection leads to destruction of CD4+T cells in the gut-associated lymphoid tissue (GALT) and promotes a decline in mechanical barrier functions of the gut mucosa, and the subsequent translocation of microbial products from the gastrointestinal tract to systemic circulation. The gut mucosal immune system is not completely restored by cART, and the resultant microbial translocation may contribute to chronic inflammation, inadequate CD4 T-cell recovery, and increased rates of serious non-AIDS events. Many studies have revealed strong and characteristic compositional differences in gut microbiota between individuals with HIV infection and seronegative controls. So far, several probiotic organisms have shown the ability to enhance intestinal epithelial barrier functions, reduce inflammation, and support effective Th-1 responses. Probiotics mainly stimulates polymeric IgA secretion, avoid bacterial overgrowth and their translocation, and produce a self-limited inflammatory response through development of regulatory T (Treg) cells by anti-inflammatory cytokine production. Therefore, we design a prospective, randomized, double-blind, placebo-controlled study to determine whether the use of a probiotic can expand beneficial microbiota that aid in decreasing bacterial translocation and pro-inflammatory cytokine production, thereby improving immune functions in HIV-infected subjects. Participants in the intervention group will receive oral probiotic containing 3 billion Bifidobacterium and 1 billion Lactobacillus once daily, while those in the placebo group will take placebo which contains no probiotic but has the same flavor and characteristics as the probiotic product.. Gut bacterial community diversity and composition, immune recovery and activation in peripheral plasma, plasma levels of gut damage, microbial translocation and inflammation at baseline and after 12 months of receiving intervention will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old;
* Documented HIV infection;
* No history of gastrointestinal diseases;
* Good adherence and promise to follow-up;
* Ability to provide informed consent.

Exclusion Criteria:

* Administration of antibiotics, probiotics, or prebiotics or experience of diarrhea within the previous 3 months;
* Administration of anti-inflammatory drugs, corticosteroids, immunosuppressive drugs, immunomodulator within the previous 3 months;
* Severe organ dysfunction;
* Pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from the Department of Infectious Diseases, Peking Union Medical College Hospital, Beijing, China. All participants are Chinese and meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Gut bacterial community diversity and composition | Change from baseline to 1 year after antiretroviral therapy
  Microbiota profiling are performed on fecal samples from each subjects, and 8-10 participants receive gastrointestinal endoscope according to their willingness

SECONDARY OUTCOMES:
Absolute CD4+ T-cell and CD8+ T-cell counts in peripheral plasma | Change from baseline to 1 year after antiretroviral therapy
  CD4+ and CD8+ T cells are analyzed by flow cytometry
The level of T cell activation and different immunophenotype in peripheral plasma | Change from baseline to 1 year after antiretroviral therapy
  CD38+HLA-DR+, CD8+CD28+ T cell subsets are analyzed by flow cytometry
Plasma levels of inflammation and coagulation markers | Change from baseline to 1 year after antiretroviral therapy
  Levels of IL-8, IL-1β, IL-6, CRP, TNF-α and D-dimer
Plasma levels of microbial translocation and monocyte activation markers | Change from baseline to 1 year after antiretroviral therapy
  Levels of I-FABP, LPS, LBP, sCD14, sCD40L, and IDO
Metabolic measurements from blood plasma | Change from baseline to 1 year after antiretroviral therapy
  Levels of vitamin D, glucose and insulin, and lipid profiling
Feasibility, safety, tolerability, adherence, and acceptability of study product and procedures | Change from baseline to 1 year after antiretroviral therapy
  Based on patients' description and intervention-related adverse events
HIV RNA | Change from baseline to 1 year after antiretroviral therapy
  HIV-RNA is detected by Roche assay with the limit of 20 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Wei LYU, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No